CLINICAL TRIAL: NCT03558555
Title: Comparative Efficacy of Intravenous Acetaminophen vs. Oral Acetaminophen in Ambulatory Surgery
Brief Title: Determine the Clinical Advantage of IV vs PO Acetaminophen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yan Lai (Other)
Responsible Party: Sponsor-Investigator, Yan Lai, Assistant Professor of Anesthesiology, Perioperative & Pain Medicine, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 16-1763; IF#16-1763 (Other: Icahn School of Medicine at Mount Sinai); IF#2175834 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Inguinal Hernia
Keywords: Acetaminophen; Tylenol; Intravenous versus oral
MeSH Terms: conditions — Hernia, Inguinal | interventions — Acetaminophen; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants presenting for inguinal hernia surgery are assigned to either the oral or intravenous acetaminophen group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral Acetaminophen (Active Comparator): Patients who are randomized to have oral acetaminophen will take oral acetaminophen preoperatively and receive saline intraoperatively.
  Interventions: Drug: Oral Acetaminophen; Drug: Saline
- Acetaminophen IV Soln (Active Comparator): Patients randomized to IV acetaminophen will receive IV acetaminophen after induction of general anesthesia and will take placebo pills preoperatively.
  Interventions: Drug: Acetaminophen IV Soln; Drug: Placebo Pills

INTERVENTIONS:
Drug: Acetaminophen IV Soln — 1000mg of IV acetaminophen
  Arms: Acetaminophen IV Soln
Drug: Oral Acetaminophen — oral acetaminophen 975mg pills
  Arms: Oral Acetaminophen
Drug: Placebo Pills — placebo match to acetaminophen
  Arms: Acetaminophen IV Soln
Drug: Saline — Intravenous saline
  Arms: Oral Acetaminophen

SUMMARY:
There is limited research on the clinical outcome differences between intravenous (IV) acetaminophen versus oral (PO) acetaminophen. With the costs of intravenous acetaminophen sometimes being almost 100 times the cost of PO acetaminophen, it is not only important fiscally but also clinically to differentiate the benefits of IV vs PO acetaminophen. The proposed research study is to determine the clinical advantages of IV vs PO acetaminophen during the post-operative recovery time for ambulatory surgery patients by analyzing differences in time to first opioid delivery, pain scores, and patient satisfaction.

DETAILED DESCRIPTION:
In previous literature it has been shown that compared to placebo, IV acetaminophen can improve postoperative pain scores and reduce opioid requirements. In addition, IV acetaminophen has several pharmacokinetic properties that may be beneficial when compared to acetaminophen. IV acetaminophen has been shown to achieve a more rapid and higher maximum plasma concentration as well as higher cerebrospinal fluid concentrations. Comparative effectiveness trials of IV vs PO administration have not conclusively demonstrated improved clinical outcomes despite the proposed pharmacokinetic benefits. More research needs to be conducted to determine possible clinical advantages.

ELIGIBILITY:
Inclusion Criteria:

* ASA scores I-III
* Ambulatory surgery patients
* Ages 18-75
* Surgeries requiring general anesthesia for hernia surgery

Exclusion Criteria:

* Patients with contraindications to acetaminophen (history of end organ liver dysfunction)
* Known allergy to acetaminophen
* Emergency surgery
* Patients who were not fasted
* Patients who cannot tolerate PO
* Surgery anticipated to last longer than 3 hours or requiring re-dose of acetaminophen
* Pregnancy
* Weight less than 50kg
* Chronic daily narcotic use
* Patients who's anesthetic plan requires regional anesthesia
* Patient refusal to participate or do not have capacity to provide consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Lai, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Helander EM, Webb MP, Bias M, Whang EE, Kaye AD, Urman RD. A Comparison of Multimodal Analgesic Approaches in Institutional Enhanced Recovery After Surgery Protocols for Colorectal Surgery: Pharmacological Agents. J Laparoendosc Adv Surg Tech A. 2017 Sep;27(9):903-908. doi: 10.1089/lap.2017.0338. Epub 2017 Jul 25. PMID 28742427
- [Background] Moller PL, Sindet-Pedersen S, Petersen CT, Juhl GI, Dillenschneider A, Skoglund LA. Onset of acetaminophen analgesia: comparison of oral and intravenous routes after third molar surgery. Br J Anaesth. 2005 May;94(5):642-8. doi: 10.1093/bja/aei109. Epub 2005 Mar 24. PMID 15790675
- [Background] Olbrecht VA, Ding L, Spruance K, Hossain M, Sadhasivam S, Chidambaran V. Intravenous Acetaminophen Reduces Length of Stay Via Mediation of Postoperative Opioid Consumption After Posterior Spinal Fusion in a Pediatric Cohort. Clin J Pain. 2018 Jul;34(7):593-599. doi: 10.1097/AJP.0000000000000576. PMID 29200016
- [Result] Patel A, Pai B H P, Diskina D, Reardon B, Lai YH. Comparison of clinical outcomes of acetaminophen IV vs PO in the peri-operative setting for laparoscopic inguinal hernia repair surgeries: A triple-blinded, randomized controlled trial. J Clin Anesth. 2020 May;61:109628. doi: 10.1016/j.jclinane.2019.109628. Epub 2019 Oct 25. PMID 31669049

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants presenting for laparoscopic hernia repair under general anesthesia in an ambulatory setting were recruited from July 2017 to December 2018. First enrollment in Dec 2017.
Groups:
- Oral Acetaminophen: Oral acetaminophen 975mg preoperatively and receive intravenous saline intraoperatively.
- Acetaminophen IV Soln: Acetaminophen 1000mg IV Soln after induction of general anesthesia and placebo pills preoperatively
Period: Overall Study
Arm/Group | Oral Acetaminophen | Acetaminophen IV Soln
Started | 58 | 45
Completed | 56 | 44
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Acetaminophen | Acetaminophen IV Soln | Total
Number analyzed (Participants) | 56 | 44 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.93 (13.37) | 52.52 (15.10) | 53.31 (14.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 33 | 24 | 57
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: PACU Visual Analogue Pain Scores
Description: Post-Anesthesia Care Unity (PACU) pain scores at baseline, 1 hour, and on discharge from PACU. Pain score by visual analogue score, total scale from 0 to 10 with 10 being the worse pain.
Time Frame: baseline, 1 hour, and Day 1 discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Acetaminophen | Acetaminophen IV Soln
Number analyzed (Participants) | 56 | 44
score on a scale
  Baseline | 2.13 (2.72) | 1.52 (2.44)
  1 hour | 2.88 (2.74) | 2.41 (2.21)
  Discharge from PACU, up to 2.5 hours | 1.45 (1.51) | 1.59 (1.44)
  6 hour post op | 3.82 (2.28) | 4.27 (1.74)
  24 hour post op | 3.64 (2.26) | 4.16 (1.83)

2. Primary Outcome: Total MME Intraoperatively
Description: Total Morphine Milligram Equivalent (MME) use intraoperatively
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Oral Acetaminophen | Acetaminophen IV Soln
Number analyzed (Participants) | 56 | 44
MME | 63.75 (21.33) | 57.24 (29.20)

3. Primary Outcome: Total Narcotic Use in PACU.
Description: Total narcotic use in PACU expressed in total morphine milligram equivalents (MME)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Oral Acetaminophen | Acetaminophen IV Soln
Number analyzed (Participants) | 56 | 44
MME | 11.33 (17.10) | 9.83 (11.99)

4. Secondary Outcome: PACU Length of Stay
Description: Time in PACU
Time Frame: up to 24 hours after PACU arrival
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Oral Acetaminophen | Acetaminophen IV Soln
Number analyzed (Participants) | 56 | 44
minutes | 82.93 (55.79) | 64.05 (33.13)

5. Secondary Outcome: Patient Reported Total Narcotic Use Post-discharge
Description: home opiod use
Time Frame: average 7 days
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Oral Acetaminophen | Acetaminophen IV Soln
Number analyzed (Participants) | 56 | 44
MME | 14.06 (14.02) | 17.56 (17.42)

6. Secondary Outcome: Patient Satisfaction.
Description: Patient satisfaction total scale from 1 to 10, with higher score indicating more satisfaction
Time Frame: 7 days post surgery
Population: one missing survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Acetaminophen | Acetaminophen IV Soln
Number analyzed (Participants) | 56 | 43
score on a scale | 5.05 (2.18) | 6.20 (3.01)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Oral Acetaminophen | Acetaminophen IV Soln
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/44
Other Adverse Events (participants affected / at risk) | 0/56 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT03558555/Prot_SAP_000.pdf